CLINICAL TRIAL: NCT05200299
Title: mFOLFOXIRI Compared to mFOLFOX6 or CapeOx as Adjuvant Chemotherapy for Stage IIIB or Stage IIIC Colorectal Cancer: A Randomized Controlled Clinical Research
Brief Title: mFOLFOXIRI Compared to mFOLFOX6 or CapeOx as Adjuvant Chemotherapy for Stage IIIB or IIIC Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T-idea
Record Dates: First submitted 2022-01-18; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2021-06

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Stage IIIC; Stage IIIB; FOLFOXIRI
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mFOLFOXIRI adjuvant chemotherapy (Experimental): Patients will receive mFOLFOXIRI once every two weeks for 12 cycles as adjuvant chemotherapy. They can change the regimen to mFOLFOX6 or CapeOx after accepting not less than two complete chemotherapy regimen, if can not tolerate the adverse reaction of mFOLFOXIRI. Total 24 weeks.
  Interventions: Drug: mFOLFOXIRI; Drug: mFOLFOX6 OR CapeOx
- mFOLFOX6 or CapeOx adjuvant chemotherapy (Active Comparator): Patients will receive mFOLFOX6 once every two weeks for 12 cycles as adjuvant chemotherapy or CapeOx once every three weeks for 8 cycles as adjuvant chemotherapy. Total 24 weeks.
  Interventions: Drug: mFOLFOX6 OR CapeOx

INTERVENTIONS:
Drug: mFOLFOXIRI — mFOLFOXIRI (oxaliplatin 85 mg/m2, irinotecan 150-165 mg/m2, and folinic acid 400 mg/m2 followed by 5-fluorouracil 2400-2800mg/m2 as a 46-48 hour continuous infusion on day 1)
  Other Names: Oxaliplatin; Irinotecan; Leucovorin; 5-Fluorouracil
  Arms: mFOLFOXIRI adjuvant chemotherapy
Drug: mFOLFOX6 OR CapeOx — mFOLFOX6(oxaliplatin 85 mg/m2, folinic acid 400 mg/m2 followed by 5-fluorouracil 2400mg/m2 as a 46-48 hour continuous infusion on day 1)
  CapeOx(Oxaliplatin 130 mg/m2 intravenous infusion on day 1,Capecitabine 1000 mg/m2 twice daily PO for 14 days)
  Other Names: Oxaliplatin; Leucovorin; 5-Fluorouracil; Capecitabine

SUMMARY:
This study will focus on postoperative patients of stage IIIB or stage IIIC colorectal cancer. These patients will start to accept chemotherapy in 3-4 weeks after operation, these patients were randomly divided into two groups, one group will accept adjuvant chemotherapy of mFOLFOX6 or CapeOX; another group will use mFOLFOXIRI, they can change the regimen to mFOLFOX6 or CapeOx after accepting not less than two complete chemotherapy regimen, if can not tolerate the adverse reaction of mFOLFOXIRI. The efficacy and safety of adjuvant chemotherapy will be compared between the two groups. Disease-free survival, overall survival, incidence of adverse reaction of chemotherapy and postoperative quality of life will be recorded.

DETAILED DESCRIPTION:
This trial is a two-arm, open labelled, prospective, randomized phase II studies. The postoperative stage of eligible patients was stage IIIB or stage IIIC. These high risk patients will be randomly assigned, in a 1:1 ratio, to receive either mFOLFOXIRI or mFOLFOX6/CapeOx for 6 months as adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* ECOG PS 0-1
* Curative surgery (R0 resection)
* ypStage III B and ypStage III C
* No distant metastasis after surgery

Exclusion Criteria:

* any treatment before surgery including chemotherapy, radiotherapy and targeted agents.
* Previous or concurrent cancer that is distinct in primary site or histology from colon cancer within 5 years prior to randomization.
* Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment.
* Heart failure grade III/IV (NYHA-classification).
* Unresolved toxicity higher than CTCAE v.4.0 Grade 1 attributed to any prior therapy/procedure.
* Subjects with known allergy to the study drugs or to any of its excipients.
* Current or recent (within 4 weeks prior to starting study treatment) treatment of another investigational drug or participation in another investigational study.
* Breast- feeding or pregnant women
* Lack of effective contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
2-year Disease-free survival | up to 2 years
  Defined as the time from randomization to relapse or death, whichever occurred first

SECONDARY OUTCOMES:
Overall survival | up to 3 years
  Defined as the time from randomization to death from any cause
The grade of toxicity will be assessed using the NCI common toxicity criteria, version 5.0. | up to 3 years
  Safety
QLQ-C30 Quality of Life questionnaire | up to 3 years
  postoperative quality of life
Quality of Life assessed by SF-36 | up to 3 years
  postoperative quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

REFERENCES:
- [Background] Falcone A, Ricci S, Brunetti I, Pfanner E, Allegrini G, Barbara C, Crino L, Benedetti G, Evangelista W, Fanchini L, Cortesi E, Picone V, Vitello S, Chiara S, Granetto C, Porcile G, Fioretto L, Orlandini C, Andreuccetti M, Masi G; Gruppo Oncologico Nord Ovest. Phase III trial of infusional fluorouracil, leucovorin, oxaliplatin, and irinotecan (FOLFOXIRI) compared with infusional fluorouracil, leucovorin, and irinotecan (FOLFIRI) as first-line treatment for metastatic colorectal cancer: the Gruppo Oncologico Nord Ovest. J Clin Oncol. 2007 May 1;25(13):1670-6. doi: 10.1200/JCO.2006.09.0928. PMID 17470860
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Stintzing S. Management of colorectal cancer. F1000Prime Rep. 2014 Nov 4;6:108. doi: 10.12703/P6-108. eCollection 2014. PMID 25580262
- [Background] Walker R, Wood T, LeSouder E, Cleghorn M, Maganti M, MacNeill A, Quereshy FA. Comparison of two novel staging systems with the TNM system in predicting stage III colon cancer survival. J Surg Oncol. 2018 Apr;117(5):1049-1057. doi: 10.1002/jso.25009. Epub 2018 Feb 23. PMID 29473957